CLINICAL TRIAL: NCT06231914
Title: Efficacy and Safety of Fractional 1064-nm Picosecond Laser for Facial Skin Tightening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Prof. Dr., Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 981/2023
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Laxity; Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fractional 1064-nm Picosecond laser (Experimental): Fractional 1064-nm Picosecond laser for 3 sessions, at 4-week interval
  Interventions: Device: StarWalker® PQX

INTERVENTIONS:
Device: StarWalker® PQX — Third-generation ASP-powered technology for ultra performance: Highest pico power & energy, shortest pico pulse width, wide range of laser wavelengths, exceptional spot size capabilities, largest fluence spectrum for flat-top handpieces

SUMMARY:
The goal of this clinical trial is to learn the efficacy and safety of fractional 1064-nm picosecond laser for facial skin tightening. The main questions it aims to answer are:

* Efficacy of fractional 1064-nm picosecond laser for facial skin efficacy including the changes in wrinkle, nasolabial fold, skin laxity, and skin elasticity
* The changes in texture and pore volume using Antera
* The changes in bioengineering assessment: melanin index, erythema index, sebum level
* Adverse events Participants will be treated with 3 sessions of fractional 1064-nm picosecond laser (full face 4 passes, vector lines 4 passes), spaced 4 weeks apart. Follow-up visits 1, 3, and 6 months after the last treatments.

DETAILED DESCRIPTION:
The efficacy and safety of fractional 1064-nm picosecond laser for facial skin tightening in participants aged 40 to 55 years, BMI < 25 kg/m2, and have mild to moderate facial laxity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-55 years
* BMI < 25 kg/m2
* Asian
* Mild to moderate facial skin laxity using quantitative grading scale (grade 1.5-2.5)

Exclusion Criteria:

* Pregnant or lactation
* Subjects who have been treated with any kind of energy-based device 6 months prior to the inclusion
* Subjects who have been injected with botulinum toxin, filler, or platelet-rich plasma on their faces 6 months prior to the inclusion
* Active skin infections
* History of hypertrophic scars or keloids

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The changes in wrinkle. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The changes in indentation of wrinkle using Antera (mm3)
The changes in nasolabial fold. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The changes in nasolabial fold using Quantificare (mm3)
The changes in skin laxity. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The changes in skin laxity using Quantificare (mm3)
The changes in skin elasticity. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The changes in skin elasticity (R0, R2, R5) using Cutometer (%)

SECONDARY OUTCOMES:
The changes in skin texture. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The measurement will be done using Antera (mm3)
The changes in pore volume. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The measurement will be done using Antera (mm3)
The change in melanin index and erythema index. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The measurement of bioengineering assessment including melanin index and erythema index using Mexameter (%)
The change in sebum level. | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  The change in sebum production using Sebumeter (%)
Adverse events | 4 weeks after the first treatment, 4 weeks after the second treatment, during 1, 3, and 6 months after the last treatment.
  Adverse events that occurred during the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand